CLINICAL TRIAL: NCT02368353
Title: Stress in At Risk Mental State: Efficacy of Stress Management Cognitive Behavioral Therapy : a Randomized Controlled Trial
Brief Title: "Stress in At Risk Mental State: Efficacy of Stress Management Cognitive Behavioral Therapy : a Randomized Controlled Trial"
Acronym: START
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D14-P008
Record Dates: First submitted 2015-02-06; First posted 2015-02-23 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Young Subjects With at Risk Mental States
MeSH Terms: interventions — Cognitive Behavioral Therapy; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral therapy group (Experimental): weekly group stress-management CBT (SM-CBT) - 1/week 3 months
  Interventions: Other: Cognitive behavioral therapy
- Reference group (Active Comparator): weekly supportive therapy - 1/week 3 months
  Interventions: Other: Supportive therapy

INTERVENTIONS:
Other: Cognitive behavioral therapy
  Arms: Cognitive behavioral therapy group
Other: Supportive therapy
  Arms: Reference group

SUMMARY:
The first psychotic episodes are preceded by a pauci-symptomatic phase from 2 to 4 years during which the psychotic symptoms are present at a subliminal level in severity or in frequency. The clinical criteria "mental status with risk" (AR) identifies patients among whom 10 in 40 % will make a psychotic transition in the year.

Our hypothesis is that interventions to reduce reactivity to stress are effective in reducing the intensity of psychotic symptoms in subjects with prodromal psychotic symptoms. Our project is to evaluate a therapy for stress management in at risk patients, compared to a conventional monitoring, and implement a longitudinal follow-up concerning the reduction of psychotic symptoms in conjunction with other markers of stress. Nonstigmatizing, these interventions offer an alternative to antipsychotics all the more interesting since they should also reduce the risk of depression and suicide.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 to 25 years
* Help-seekers in one of the specialized clinics for adolescents or young adults 9
* Meets CAARMS criteria for 'at risk mental state' (ARMS)

Exclusion Criteria:

* situations of emergency.
* prengnancy, breast-feeding
* Forced hospitalization or individuals under legal guardianship.
* schizophrenia (DSMIV-TR criteria)
* Low IQ (<70) ,
* Mother tongue and primary educational language other than French
* Blindness, deafness, muteness, sensorimotor or language deficits
* any severe medical condition,
* Daily cannabis use in the last week
* Current depression (>20 MADRS scale)
* Substance dependence or abuse (except nicotine) for more than 5 years.
* Treatments by benzodiazépine (> 10 mg amount diazépam) or stop of less than 5 days
* Previous treatment by antipsychotics in a superior dose in more than 100 mg equivalent Chlorpromazine if at least a sequence lasted more than 12 weeks
* Treatment by antipsychotics measures > 100 mg eq. CPZactuel (superior dose in more than 100 mg equivalent Chlorpromazine) so introduced for less than three weeks
* Antidepressant treatmentsbegun for less three weeks
* Treatment by corticoids (except local treatment)
* Exclusion period of another study;
* The usual contraindications for MRI
* Absence of social insurance

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-02-13 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The score at month 6 on the "positive" psychotic dimension of the CAARMS (first subscale including delusion, hallucination and disorganized thoughts). | Month 6

SECONDARY OUTCOMES:
Score on CAARMS | Month 0
Score on CAARMS | Month 6
Score on CAARMS | Month 12
· Rate of conversion (as defined by CAARMS) | Month 6
· Rate of conversion (as defined by CAARMS) | Month 12
Score on BPRS | Month 0
Score on BPRS | Month 6
Score on BPRS | Month 12
Score on MADRS | Month 0
Score on MADRS | Month 6
Score on MADRS | Month 12
Score on YMRS | Month 0
Score on YMRS | Month 6
Score on YMRS | Month 12
Score on SOFAS | Month 0
Score on SOFAS | Month 6
Score on SOFAS | Month 12
Stress marker : saliva cortisol level | Month 0
Stress marker : saliva cortisol level | Month 6
Stress marker : saliva cortisol level | Month 12
Stress marker : telomerase activity | Month 0
Stress marker : telomerase activity | Month 6
Stress marker : telomerase activity | Month 12
Stress marker : epigenetic markers | Month 0
Stress marker : epigenetic markers | Month 6
Stress marker : epigenetic markers | Month 12
Stress marker : genetic variants that modulate stress response | Month 0
Stress marker : genetic variants that modulate stress response | Month 6
Stress marker : genetic variants that modulate stress response | Month 12
Stress marker : hippocampal volume | Month 0
Stress marker : hippocampal volume | Month 12
Performance score on autobiographic memory | Month 0
Performance score on autobiographic memory | Month 12
Performance score on sense of self tasks | Month 0
Performance score on sense of self tasks | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France